CLINICAL TRIAL: NCT06446570
Title: Phase II Study of Durvalumab +/- Tremelimumab in Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Phase II Study of Durvalumab(MEDI4736) + Tremelimumab in Pulmonary Sarcomatoid Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-16-12012
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: HNSCC; Head and Neck Neoplasms
Keywords: biomarker driven umbrella trial; Durvalumab + Tremelimumab Combination Treatment
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab, tremelimumab (Experimental): Durvalumab is a human immunoglobulin (Ig) G1 kappa (IgG1κ) monoclonal antibody (mAb) that blocks the interaction of PD-L1 with PD-1 on T-cells and CD80 on immune cells and is engineered to reduce antibody-dependent cell-mediated cytotoxicity.(IV class)
  Tremelimumab is specific for human CTLA-4; cluster of differentiation a cell surface receptor that is expressed primarily on activated T cells and acts to inhibit their activation.(IV class)
  Interventions: Drug: Durvalumab,Tremelimumab

INTERVENTIONS:
Drug: Durvalumab,Tremelimumab — Durvalumab: 1.5g Q4W plusTremelimumab: 75mg Q4W up to 4cycle then Durvalumab 750mg Q2W, till PD or unacceptable toxicity.
  Other Names: Experimental group

SUMMARY:
Phase II study of Durvalumab+/- Tremelimumab in patients with recurred metastatic head and neck squamous cell carcinoma

DETAILED DESCRIPTION:
Open, multicenter, single arm, phase II, biomarker driven umbrella trial for head and neck squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* 1. Recurrent or metastatic HNSCC, regardless of PD-L1 or HPV status 2. Age ≥20 3. ECOG PS 0-1 4. Ineligibility for local therapy (surgery or radiotherapy) 5. Prior palliative chemotherapy including platinum-based chemotherapy. When recurred within 6 months of definitive/neoadjuvant/adjuvant chemo- or chemoradiation, the chemotherapy is considered a line of therapy 6. At least one measurable lesion by RECIST ver 1.1 7. Adequate organ function for treatment
* Absolute neutrophil count (ANC) ≥1000 cells/mm3
* Hemoglobin: ≥ 9.0 g/dL
* Platelets ≥100,000 cells/mm3
* Estimated creatinine clearance ≥40 mL/min, or serum creatinine <1.5 x institution upper limit of normal
* Bilirubin ≤1.5 x upper limit of normal (ULN)
* AST (SGOT) ≤2.5 x ULN (5.0 x ULN if hepatic metastases)
* ALT (SGPT) ≤2.5 x ULN (5.0 x ULN if hepatic metastases) 8. 12-Lead electrocardiogram (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention 9. The patient has provided signed informed consent

Exclusion Criteria:

* 1. Previous treatment with PD-1 or PDL-1 inhibitors 2. Nasopharyngeal carcinoma 3. Cytotoxic chemotherapy within 3 weeks of study entry; immunotherapy or investigational drug within 5 half-lives of study entry 4. Any major operation or irradiation within 4 weeks of baseline disease assessment. Palliative radiation is allowed 5. Symptomatic brain metastasis 6. Patients with known interstitial lung disease 7. Patients with uncontrolled or significant cardiovascular disease 8. Previous or concurrent malignancy (except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, thyroid cancer treated curatively) without evidence of recurrence for at least 3 years prior to study entry.

  9. Pregnant or breast-feeding women 10. Systemic immunosuppressive therapy 11. Active autoimmune disease 12. Patient who have an active systemic fungal and/or known viral infection (for example, human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C antibodies) (inactive HBV carrier with adequate prophylactic antiviral agent can be enrolled) 13. Body weight <30kg

  14. Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) | 24months
  RECIST1.1

SECONDARY OUTCOMES:
•Progression-Free Survival (PFS) | 24months
  Disease progression is assessed by RECIST 1.1.
•Overall Survival (OS) | 24months
  Overall Survival is defined as the time from first dose to death due to any cause. Through the follow-up within 30 days after study completion or termination of the last subject, death and date of death will be checked for subject alive during treatment period
•Toxicity | 24months
  number of patients with treatment-related AE as assessed by NCI CTCAE version 4.03
•biomarker | 24months
  NGS, nanostring technology

CONTACTS AND LOCATIONS:
Overall Officials: Bhumsuk Keam, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
anticipated as research paper